CLINICAL TRIAL: NCT05857878
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Rising Oral Doses of BI 1815368 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Well Different Doses of BI 1815368 Are Tolerated by Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1485-0002; 2023-503815-13-00 (Registry Identifier: CTIS); 2022-002278-96 (EudraCT Number)
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo
- Dose Group 1 (Experimental)
  Interventions: Drug: BI 1815368
- Dose Group 2 (Experimental)
  Interventions: Drug: BI 1815368
- Dose Group 3 (Experimental)
  Interventions: Drug: BI 1815368
- Dose Group 4 (Experimental)
  Interventions: Drug: BI 1815368
- Dose Group 5 (Experimental)
  Interventions: Drug: BI 1815368
- Dose Group 6 (Experimental)
  Interventions: Drug: BI 1815368

INTERVENTIONS:
Drug: BI 1815368 — BI 1815368
  Arms: Dose Group 1; Dose Group 2; Dose Group 3; Dose Group 4; Dose Group 5; Dose Group 6
Drug: Matching placebo — Matching placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This trial aims to investigate safety, tolerability, and pharmacokinetics following multiple rising doses of BI 1815368 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests.
* Age of 18 to 55 years (inclusive).
* Body mass index (BMI) of 19 to 29.9 kg/m2 (inclusive).
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator.
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm).
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair).
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders.
* History of relevant orthostatic hypotension, fainting spells, or blackouts. Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients treated who experience treatment-emergent adverse event assessed as drug-related by the investigator | Up to 29 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 1815368 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | Up to 16 days
Minimum concentration of BI 1815368 in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | Up to 16 days
Maximum measured concentration of BI 1815368 in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | Up to 16 days

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com